CLINICAL TRIAL: NCT00032721
Title: The Use of Reiki for Patients With Advanced AIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R21AT001012-01 (NIH)
Record Dates: First submitted 2002-03-29; First posted 2002-04-01 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: complementary therapies; Alternative medicine; Complementary and alternative medicine; Subtle energy therapy; Reiki; HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Therapeutic Touch

INTERVENTIONS:
Procedure: Reiki; Subtle energy therapy

SUMMARY:
This study will investigate the use of Reiki, an energy-based complementary and alternative medicine (CAM) intervention, as an approach to improve well-being for patients with advanced AIDS, and evaluate its effects on dimensions of well-being and quality of life.

DETAILED DESCRIPTION:
This study will investigate the use of Reiki, an energy-based complementary and alternative medicine (CAM) intervention, as an approach to improve well being for patients with advanced AIDS, and evaluate its effects on dimensions of well being and quality of life. The study is a two-group comparison between participants receiving Reiki plus usual medical care (treatment) and participants receiving usual medical care only (control).

One hundred and forty-six patients with advanced AIDS will be enrolled and randomized into the two groups. Patients in the intervention (Reiki) group will receive a total of three one-hour Reiki sessions over a period of 6 weeks. Participants in both the intervention and control groups will be assessed at two times during the study period using repeated measures. We will investigate and compare changes in participants' anxiety, depression, pain, quality of life, and spiritual well being at the end of the intervention period. This is the first part of a longer-term research agenda to examine the use and effectiveness of complementary and alternative medicines for patients with advanced disease. We plan to examine one clinical context in which Reiki is currently provided. It is important to design studies that respect both the context of care and the practitioner-client relationship-elements essential to an understanding of the philosophy and delivery of CAM such as Reiki, and at the same time endeavor to outline a systematic approach to the study of CAM.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of advanced AIDS, defined as: CD4 count of less than 200 during the past 12 months;
* On HAART for at least 6 months;
* Over age 18;
* Decisionally capable of providing informed consent.

Exclusion Criteria:

* Not capable of providing informed consent because of psychiatric limitations, e.g. active psychosis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146
Dates: Start 2002-03; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Gala True, PhD, Principal Investigator — Albert Einstein Healthcare Network
Locations (2):
- United States (2):
  - Temple University, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania